CLINICAL TRIAL: NCT04434118
Title: Anti-rheumatic Drug Use and Risk of COVID-19 Infection in Rheumatoid Arthritis Patients: A Retrospective, Case-control Study
Brief Title: Anti-rheumatic Drug Use and Risk of COVID-19 Infection in Rheumatoid Arthritis Patients
Status: Withdrawn | Type: Observational
Why Stopped: Institutional Issue
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Mahmoud Samy Abdallah, Lecturer of Clinical Pharmacy, PhD., Sadat City University
Other Study IDs: IRB: RC-5-2020
Record Dates: First submitted 2020-06-13; First posted 2020-06-16 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis; COVID
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rheumatoid Arthritis with COVID-19
  Interventions: Drug: Traditional antirheumatic drugs
- Rheumatoid Arthritis without COVID-19
  Interventions: Drug: Traditional antirheumatic drugs

INTERVENTIONS:
Drug: Traditional antirheumatic drugs — Hydroxychloroqine, Methotrexate, Glucocorticoids, Leflunomide, and Sulphasalazine

SUMMARY:
Rheumatoid arthritis (RA) patients have an underlying immune deficiency and typically treated with immunosuppressive drugs, which may increase the risk of COVID-19 infection. Hydroxychloroquine (HCQ) has been found to possess antiviral activity against COVID-19. Thus, the aim of this study to investigate the ability of HCQ to reduce the risk of COVID-19 among RA patients.

ELIGIBILITY:
Inclusion Criteria:

- Data of all definite cases of RA were collected and reviewed from complete medical records of patients by a team that included 2 trained physicians using a pretested data collection form.

Exclusion Criteria:

* The exclusion criteria were included incomplete medical records or those with difficulty to communicate with the patients.
* Patients with acute lethal organ injury (e.g., acute myocardial infarction, acute coronary syndrome, acute pulmonary embolism, or acute stroke)
* Patients with decompensated or end stage chronic organ dysfunction (e.g., decompensated cirrhosis, decompensated chronic renal insufficiency, or severe congestive heart failure), diabetes mellitus, data of pregnant females, acquired immune deficiency syndrome (aids), and leukemia or other malignancies.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients fulfilling 2010 ACR-EULAR classification criteria for RA
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
The risk of COVID-19 infection among RA patients | 12 week
  Realtion between hydroxychloroquine use and COVID-19 infection

SECONDARY OUTCOMES:
The incidence of hospitalization for Covid-19 patients. | 12 week
  Number of cases and number of hospitalization days

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP